CLINICAL TRIAL: NCT01088451
Title: Joint Application of Human Insulin and Rapid Insulin Analogue in Control of Postprandial Glycemia
Acronym: CPIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: David Neumann/Principal Investigator, University Hospital Hradec Králové
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200912S24; MZO00179906-01 (Other Grant/Funding Number: University Hospital Hradec Králové)
Record Dates: First submitted 2010-02-11; First posted 2010-03-17 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Prandial Glycemia; Rapid Acting Insulin Analogue; Human Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Combined prandial insulin therapy (CPIT) — Combined prandial insulin therapy (CPIT) applies individual combination of rapid insulin analogue and human insulin according subject's individual estimation of the type of carbohydrates in concrete mixed-meal, based on thorough education. In this study subjects use two applicators, giving two injections before main meals as per basal-bolus therapy. Insulin aspart (Novorapid, Novo Nordisk) and human insulin (Actrapid, Novo Nordisk) are used.

SUMMARY:
Postprandial glycemic control is essential for diabetes compensation. Insulin pump therapy control blood glucose released in response to both high and low glycemic index carbohydrates in a mixed diet using normal, square and dual-wave boluses. The investigators hypothesize a mixture of rapid insulin analogue and human insulin has the same effect.

This pilot prospective cohort study replaces basal-bolus therapy of diabetic subjects by combined prandial application of insulin aspart and human insulin. Mixed-meals with high, both high and low and low glycemic index carbohydrates are covered by 3:1, 1:1 and 1:3 ratios of analogue to human insulin mixture. Subjects are followed by continuous glucose monitor for six days (Phase One), changing between the experimental or their standard protocol for insulin injection on consecutive days. The outcome was measured by comparing average glycemia and areas under the curve of sample meals, which are doughnut, pizza and mixed vegetable salad. The next three-to-four week period of therapy was evaluated by glycated hemoglobin before and after the intervention (Phase Two).

Expected outcomes are postprandial and complex improvement of diabetes control, similarly to the insulin pump therapy.

ELIGIBILITY:
Inclusion criteria

* pubertal children, adolescents, young adults able to follow instructions, regardless of their long-time compliance
* willing to undertake a prandial application of two kinds of insulin using two standard insulin applicators.
* willing to complete detailed meal, insulin and/or combination insulin and hypoglycemia diary throughout the study.

Exclusion criteria:

* acute illness and celiac disease, but not euthyroid autoimmune thyroiditis, defined as thyroid stimulating hormone (TSH)<4 mIU/l.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-03 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Differences in mean blood glucose concentrations and the pattern of fluctuation on control and study days; and changes in the glycated hemoglobin A1c after the study period. Occurrence of side effects especially hypoglycemic episodes. | one month

SECONDARY OUTCOMES:
The difference in postprandial areas under the curve when comparing conventional therapy and experimental combined prandial insulin therapy in the 5 to 6 hours following meal ingestion, taking into account the glycemic index profile of the meal. | one month

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Králové, Hradec Králové, Czechia

REFERENCES:
- [Background] Monnier L, Lapinski H, Colette C. Contributions of fasting and postprandial plasma glucose increments to the overall diurnal hyperglycemia of type 2 diabetic patients: variations with increasing levels of HbA(1c). Diabetes Care. 2003 Mar;26(3):881-5. doi: 10.2337/diacare.26.3.881. PMID 12610053
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Franceschi S, Hamidi M, Marchie A, Jenkins AL, Axelsen M. Glycemic index: overview of implications in health and disease. Am J Clin Nutr. 2002 Jul;76(1):266S-73S. doi: 10.1093/ajcn/76/1.266S. PMID 12081850
- [Background] Flint A, Moller BK, Raben A, Pedersen D, Tetens I, Holst JJ, Astrup A. The use of glycaemic index tables to predict glycaemic index of composite breakfast meals. Br J Nutr. 2004 Jun;91(6):979-89. doi: 10.1079/bjn20041124. PMID 15182401
- [Background] Monro J. Redefining the glycemic index for dietary management of postprandial glycemia. J Nutr. 2003 Dec;133(12):4256-8. doi: 10.1093/jn/133.12.4256. PMID 14652382
- [Background] Brouns F, Bjorck I, Frayn KN, Gibbs AL, Lang V, Slama G, Wolever TM. Glycaemic index methodology. Nutr Res Rev. 2005 Jun;18(1):145-71. doi: 10.1079/NRR2005100. PMID 19079901
- [Background] Axelsen M, Wesslau C, Lonnroth P, Arvidsson Lenner R, Smith U. Bedtime uncooked cornstarch supplement prevents nocturnal hypoglycaemia in intensively treated type 1 diabetes subjects. J Intern Med. 1999 Mar;245(3):229-36. doi: 10.1046/j.1365-2796.1999.00432.x. PMID 10205584
- [Background] O'Connell MA, Gilbertson HR, Donath SM, Cameron FJ. Optimizing postprandial glycemia in pediatric patients with type 1 diabetes using insulin pump therapy: impact of glycemic index and prandial bolus type. Diabetes Care. 2008 Aug;31(8):1491-5. doi: 10.2337/dc08-0306. Epub 2008 May 28. PMID 18509207
- [Background] Pankowska E, Szypowska A, Lipka M, Szpotanska M, Blazik M, Groele L. Application of novel dual wave meal bolus and its impact on glycated hemoglobin A1c level in children with type 1 diabetes. Pediatr Diabetes. 2009 Aug;10(5):298-303. doi: 10.1111/j.1399-5448.2008.00471.x. Epub 2008 Oct 20. PMID 19175902
- [Background] Report of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Diabetes Care. 1997 Jul;20(7):1183-97. doi: 10.2337/diacare.20.7.1183. No abstract available. PMID 9203460
- [Background] Bowden SA, Duck MM, Hoffman RP. Young children (<5 yr) and adolescents (>12 yr) with type 1 diabetes mellitus have low rate of partial remission: diabetic ketoacidosis is an important risk factor. Pediatr Diabetes. 2008 Jun;9(3 Pt 1):197-201. doi: 10.1111/j.1399-5448.2008.00376.x. PMID 18547233
- [Background] Workgroup on Hypoglycemia, American Diabetes Association. Defining and reporting hypoglycemia in diabetes: a report from the American Diabetes Association Workgroup on Hypoglycemia. Diabetes Care. 2005 May;28(5):1245-9. doi: 10.2337/diacare.28.5.1245. No abstract available. PMID 15855602
- [Background] Foster-Powell K, Holt SH, Brand-Miller JC. International table of glycemic index and glycemic load values: 2002. Am J Clin Nutr. 2002 Jul;76(1):5-56. doi: 10.1093/ajcn/76.1.5. PMID 12081815
- [Background] Hirsch IB. Insulin analogues. N Engl J Med. 2005 Jan 13;352(2):174-83. doi: 10.1056/NEJMra040832. No abstract available. PMID 15647580
- [Background] Pickup J, Mattock M, Kerry S. Glycaemic control with continuous subcutaneous insulin infusion compared with intensive insulin injections in patients with type 1 diabetes: meta-analysis of randomised controlled trials. BMJ. 2002 Mar 23;324(7339):705. doi: 10.1136/bmj.324.7339.705. PMID 11909787